CLINICAL TRIAL: NCT06554561
Title: The Safety and Efficacy of Pomadomide in Combination With Rituximab and Methotrexate for Newly-diagnosed Primary Central Nervous System Lymphoma : A Prospective, Multicenter, Phase I/II Study
Brief Title: A Study of Pomadomide in Combination With Rituximab and Methotrexate for Newly-diagnosed Primary Central Nervous System Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IR2024280
Record Dates: First submitted 2024-08-07; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: PCNSL
Keywords: PCNSL; Pomadomide; Rituximab; Methotrexate
MeSH Terms: interventions — pomalidomide; Rituximab; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PRM treatment (Experimental): Experimental arm will be treated with PRM regimen (pomadomide in combination with rituximab and methotrexate) for 4 cycles as initiate induction. If the patients achieved complete remission（CR）or partial remission（PR）, They would be consolidated by autologous transplantation consolidation regimen or the original regimen for additional 2 courses, and then were given pomadomide maintenance therapy for 12 cycles.
  Interventions: Drug: Pomalidomide; Drug: Rituximab; Drug: Methotrexate

INTERVENTIONS:
Drug: Pomalidomide — 3-5mg d1-d14 for 4-6 cycles, every 21 days as induction/consolidation chemotherapy, Then 3-5mg d1-d14 for 12 cycles, every 28 days as maintenance treatment.
Drug: Rituximab — 375mg/m2 intravenous infusion d1, every 3 weeks for 1 cycle, 4-6 cycles will be prescribed.
Drug: Methotrexate — 3.5g/m2 intravenous infusion for 4 hours in d1, every 21 days for 1 cycle, 4-6 cycles will be prescribed.

SUMMARY:
This is a prospective, multicenter, single-arm, open Phase Ib/II clinical study to explore the safety and efficacy of pomadomide in combination with rituximab and methotrexate (RPM) in newly diagnosed primary central nervous system lymphoma (PCNSL) subjects. The Phase I study is a dose escalation study, in which rituximab and methotrexate are fixed doses, and pomadomide is set into 3 dose groups: 3mg/d, 4mg/d and 5mg/d. In strict accordance with the "3+3" dose escalation principle, 3-6 subjects are to be recruited in each dose group, and each subject is to be observed for 1 cycle after treatment to determine MTD. Phase II study: RP2D is planned to be determined based on the Phase Ib study, with an additional 25 active participants enrolled to further evaluate efficacy and safety. Subjects with initial treatment of PCNSL who met the inclusion/exclusion criteria were screened, and after signing the informed consent letter, they received 4 courses of PRM regimen. The patients achieving CR or PR were consolidated by autologous transplantation consolidation regimen or the original regimen for 2 courses, and then were given pomadomide maintenance therapy for 12 cycles. Follow-ups should be taken up to the first 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed CD20+ diffuse large B-cell lymphoma (DLBCL).
* The lesions were confined to the central nervous system, including the brain, spinal cord, eyes and meninges.
* Through physical examination, imaging examination (including CT, MRI, PET-CT, etc.) and bone marrow puncture examination, it was confirmed that no parts other than the central nervous system were involved.
* Patients who have not previously received chemotherapy or radiotherapy (except those with dexamethasone less than 10mg/ day (or equivalent dose) and duration less than 5 days).
* Aged between 18 and 75 (inclusive).
* Eastern Cooperative Oncology Group performance status 0 to 3.
* Measurable disease was defined as at least ≥1.0cm in short-diameter by enhanced MRI.
* Life expectancy of ≥ 3 months (in the opinion of the investigator).
* Participants must be able to understand and be willing to sign a written informed consent document.
* Participants can follow up on schedule, communicate well with the investigator and complete the trial according to the trial regulations.
* Women of reproductive potential must agree to use highly effective methods of birth control during the period of therapy and for 6 months after the last dose of the study drug. Men who are sexually active must agree to use highly effective contraception during the period of therapy and for 6 months after the last dose.

Exclusion Criteria:

* Have systemic lymphoma disease.
* Previous systemic or local treatment such as chemotherapy and/or radiotherapy and/or hematopoietic stem cell transplantation.
* Previous or concurrent history of other malignant tumors requiring active therapy.
* Chronic or currently active infectious diseases requiring systemic antibiotic, antifungal, or antiviral treatment (except EBV infections).
* Accompanied by uncontrolled cardiovascular and cerebrovascular diseases, bleeding diseases, thrombotic diseases, connective tissue diseases and other diseases.
* Patients with other uncontrolled diseases that the researchers deemed unsuitable for inclusion.
* Laboratory test values at screening (unless due to lymphoma) : White blood cell count < 3.5×109/L, neutrophils <1.5×109/L, platelets <80×109/L, hemoglobin <100g/L, ALT or AST 2.5 times higher than the upper limit of normal, bilirubin 1.5 times higher than the upper limit of normal, creatinine level 1.5 times higher than the upper limit of normal.
* Presence of active hepatitis B virus(HBV) infection (HBsAg positive and HBV-DNA≥ 104), hepatitis C virus(HCV) infection, acquired and congenital immunodeficiency diseases include but not limited to HIV. HbsAg positive patients need to check HBV-DNA < 10^4 to be enrolled. In addition, if HBsAg is negative but HBcAb is positive (regardless of HBsAb status), HBV-DNA testing is also required, and HBV-DNA results < 10^4 are required to be enrolled and continue treatment and monitoring of HBV-DNA. HCV antibody positive patients need to check HCV-RNA quantitative DNA < 10^3 to be enrolled.
* Pregnant or lactating women.
* Those with a history of drug use or abuse were asked.
* Patients with mental illness or other patients known or suspected to be unable to fully comply with the study protocol.
* Known allergy to the investigational drug or its related ingredients.
* Patients are unable to swallow capsules or suffer from diseases or conditions that severely affect gastrointestinal function, such as malabsorption syndrome, removal of the stomach or small intestine, or complete intestinal obstruction.
* Patients who cannot withstand enhanced MRI.
* Participants considered unsuitable for this clinical trial due to various other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2024-08-31 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
MTD | 21days
  MTD of pomalidomide when given in combination with rituximab and methotrexate determined by dose-limiting toxicities graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0
Objective response rate(ORR) | 4 cycles of threatment
  The objective response rate is defined as the proportion of patients with a response of complete response(CR) or partial response(PR).

SECONDARY OUTCOMES:
Progression free survival | Time from registration to progression or death due to PCNSL, assessed up to 2 years
  From date of patients sign informed consent until the date of progression or death or the date of last follow-up time, whichever came first, assessed up to 3 years
Overall survival | Time from registration to death due to any cause, assessed up to 3 years
  From date of patients sign informed consent until the date of progression or death or the date of last follow-up time, whichever came first, assessed up to 3 years

OTHER OUTCOMES:
pomalidomide levels in the CNS | Up to day 3 of course 2
  Based on pomalidomide levels in CSF at different time points
pomalidomide levels in the Blood | Up to day 3 of course 2
  Based on pomalidomide levels in blood at different time points

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No